CLINICAL TRIAL: NCT05831332
Title: Safety and Efficacy of the BTL-785F Device for Non-invasive Reduction of Submental Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTBG200
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BTL-785-7 Treatment (Experimental): Treatment with the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat.
  Interventions: Device: BTL-785-7

INTERVENTIONS:
Device: BTL-785-7 — Treatment with the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive reduction of submental fat and skin laxity treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of submental fat
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible excess fat in submentum as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)1
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Nerve insensitivity (sensitivity disorders) to heat in the treatment area
* Varicose veins, pronounced edemas1
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use fat reduction, anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Electroanalgesia without exact diagnosis of pain etiology
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Change of submental fat thickness | 6 months
  To gather clinical evidence that BTL-785F system equipped with BTL-785-7 applicator is able to provide reduction of submental fat thickness.

SECONDARY OUTCOMES:
Evaluation the effect on submental skin laxity | 6 months
  To gather clinical evidence that BTL-785F system equipped with BTL-785-7 applicator is able to provide improved skin laxity in the submental area.
Evaluation the safety of the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat. | 6 months
  To evaluate the safety of the BTL-785F device with the BTL-785-7 applicator for non-invasive reduction of submental fat through monitoring of adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for specialized medical care - Individual dermatological practice Dr. Mariya Genova, Plovdiv, Bulgaria